CLINICAL TRIAL: NCT03599297
Title: Evaluation of Efficacy and Safety Profile of Bilateral Synchronous Simultaneous Stone Surgery for Kidney Stones
Brief Title: Bilateral Synchronous Simultaneous Stone Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAR.UAD.003
Record Dates: First submitted 2018-06-04; First posted 2018-07-26 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Kidney Calculi; Nephrolithotomy, Percutaneous; Ureteroscopy
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bilateral synchronous simultaneous stone surgery (Experimental): Patients who will be operated for kidney stones at both their kidneys in a single surgery session will be included in the study. Patients will undergo percutaneous nephrolithotomy for one side and flexible ureteroscopy for the other side.
  Interventions: Procedure: Bilateral synchronous simultaneous stone surgery

INTERVENTIONS:
Procedure: Bilateral synchronous simultaneous stone surgery — Patients undergoing Bilateral synchronous simultaneous stone surgery (one kidney undergoing percutaneous nephrolithotomy, other kidney undergoing ureteroscopy at the same time in a single patient)

SUMMARY:
Advancements in technology and endourological armamentarium provides multiple surgical options for complicated stone patients. To avoid multiple operations and shorten the total operation durations, bilateral synchronous simultaneous stone surgery (BSSSS) has been popularized in recent years.

Our aim is to evaluate the preliminary outcomes of BSSSS in patients undergoing supine percutaneous nephrolithotomy (PCNL) and retrograde intrarenal surgery (RIRS).

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for kidney stone surgery according to European Association Urology, Urolithiasis guidelines
* patients with bilateral kidney stones

Exclusion Criteria:

* none

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Stone free rate | at the 24th hour of the surgery
  stone free status is decided according to both the immediate evaluation of the endoscopic view at the end of the operation and the post operative imaging with kidney, ureter, bladder X-ray at the 24th hour of the surgery

SECONDARY OUTCOMES:
Complications | at the 1st week of surgery
  Complications are assessed according to Clavien Dindo classification
Post operative urinary diversion | at the 24th hour of surgery
  evaluation of patients whether they have a nephrostomy or a ureteral stent at the end of the operation
Radiation exposure | At 1st hour of surgery
  The cumulative fluoroscopy dose that was emitted during surgery
Hemoglobin level change | from baseline to 24th hour of surgery
  The amount of hemoglobin drop during and after surgery
Hospital stay | will be assessed through completion of study, an average of 1 year.
  The amount of days that the patient stayed at the hospital
Residual stone | at the 24th hour of surgery
  The diameter of the stones that couldn't be retracted

CONTACTS AND LOCATIONS:
Overall Officials: Yiloren Tanidir, Ass. Prof., Principal Investigator — Marmara University, School of Medicine, Department of Urology
Locations (1):
- Marmara University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data will not be shared.